CLINICAL TRIAL: NCT04337164
Title: Observational Tomodensitometric Study of the Anatomical Landmarks Depth Required to Perform Femoral Nerve Block or PENG Block. The Tomo-PENG Study.
Brief Title: Radiological Study of PENG Block Depth
Acronym: Tomo-PENG
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire de Besancon (Other)
Responsible Party: Sponsor
Other Study IDs: 2020-495
Record Dates: First submitted 2020-03-31; First posted 2020-04-07 (Actual); Last update posted 2020-12-21 (Actual); Status verified 2020-12

CONDITIONS: Regional Anesthesia; Computed Tomography; Anatomical Description
Keywords: PENG block

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This study evaluates the depth of anatomical landmarks required in regional anaesthesia to perform either Femoral Nerve Block or PENG Block.

Measures will be performed on abdominal and pelvic computed tomography as part of daily routine patient care.

DETAILED DESCRIPTION:
PENG Block is a new approach in regional anesthesia for hip surgery. The anatomical landmarks used to perform PENG Block are deeper than those for Femoral Nerve Block. Nevertheless, depth required for PENG Block is not yet evaluated since it may vary between patients.

Daily routine abdominal and pelvic computed tomography allow such anatomical description.

ELIGIBILITY:
Inclusion Criteria:

* All adult patients who have had a CT scan including visualization of the pelvis and who have expressed no opposition

Exclusion Criteria:

* pregnancy
* Subject presenting a pathology likely to modify the anatomical landmarks studied: ie pelvic fracture, psoas haematoma, previous pelvic surgery or hip prosthesis or femoral bypass

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who had a CT scan in a single institution
Sampling Method: Non-Probability Sample
Enrollment: 101 (Actual)
Dates: Start 2020-04-08 (Actual); Primary Completion 2020-07-10 (Actual); Study Completion 2020-07-10 (Actual)

PRIMARY OUTCOMES:
PENG Block depth | 1 hour after radiological examination
  Measure of puncture depth required to achieve a PENG Block on CT Scann images

SECONDARY OUTCOMES:
Femoral Nerve Block depth | 1 hour after radiological examination
  Measure of puncture depth required to achieve a Femoral Nerve Block on CT Scann images
puncture angle needed | 1 hour after radiological examination
  Measure of puncture angle that would be required to achieve a PENG Block depth on CT Scann images
needle length needed | 1 hour after radiological examination
  Measure of needle length that would be required to achieve a PENG Block depth on CT Scann images

CONTACTS AND LOCATIONS:
Locations (1):
- Centre Hospitalier Universitaire, Besançon, France

IPD SHARING:
Plan to Share IPD: Undecided
In accordance with future institutional decisions